CLINICAL TRIAL: NCT06676501
Title: A Study to Evaluate the Safety and Efficacy of Staged Bilateral Magnetic Resonance-Guided Focused Ultrasound Thalamotomy for the Treatment of Essential Tremor
Acronym: ET-Bi-MRgFUS
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Longsheng Pan, Professor, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 301ET-2
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Last update posted 2024-11-06 (Actual); Status verified 2024-11

CONDITIONS: Essential Tremor; Essential Tremor, Movement Disorders
Keywords: MRgFUS; focused ultrasound; Thalamotomy
MeSH Terms: conditions — Essential Tremor; Movement Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ExAblate Treatment (Experimental): Participants will undergo a thalamotomy contralateral to their previous treatment with MRgFUS
  Interventions: Procedure: ExAblate

INTERVENTIONS:
Procedure: ExAblate — Transcranial focused ultrasound thalamotomy

SUMMARY:
The objective of this prospective, single-arm, open-label study is to asses the safety and efficacy of the staged bilateral thalamotomy using transcranial magnetic resonance guided focused ultrasound system ExAblate 4000, InSightec Ltd.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women age 22 years or older
2. Subject is able and willing to give consent and able to attend all study visits
3. Subject is diagnosed with Essential Tremor as confirmed by a movement disorder specialist
4. Subject's tremor is refractory to adequate trials of at least two medications, one of which being a first line therapy of either propranolol or primidone. An adequate medication trial is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated.
5. Subject is diagnosed with medication-refractory Essential Tremor
6. A subject who underwent an Exablate index procedure in a clinical trial or in a commercial setting at least 9 months prior to enrolling in this trial
7. Subject has a baseline CRST Part A score of 2 or above for postural or intention tremor severity in the upper extremity for the contralateral tremor side while on stable medication
8. Subject is able to communicate sensations during the Exablate thalamotomy procedure.
9. Subject has a baseline CRST Part C score of 2 or above in any one of the items (speaking, eating, drinking, hygiene, dressing, writing, working, and social activities).

Exclusion Criteria:

1. Subject experienced any non-transient neurological event or worsening following the Exablate index procedure
2. Subject has physical subscale score ≥ 16.5 on the Dysphagia Handicap Index or has been diagnosed with dysphagia
3. Subject has score <22 on the Montreal Cognitive Assessment (MoCA)
4. Subject has any non-transient hemiparesis as determined by physical examination
5. Subject with clinically significant abnormal speech function as determined by a speech pathologist
6. Subject of childbearing potential is pregnant or breastfeeding
7. Subject with unstable cardiac status including:

   1. Unstable angina pectoris on medication
   2. documented myocardial infarction within six months of enrollment
   3. Unstable or worsening congestive heart failure
   4. History of a hemodynamically unstable cardiac arrhythmia
   5. Cardiac pacemaker
   6. Severe hypertension (diastolic BP > 100 on medication)
8. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse
9. Subject has history of abnormal systemic or intracranial bleeding, hemorrhage, or coagulopathy
10. Subject has abnormal coagulation profile: (PLT < 100,000/μl), PT (>14 sec) or PTT (>36 sec), and INR > 1.3
11. Subject receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of Exablate procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of Exablate procedure
12. Subject with cerebrovascular disease, including but not limited to, intracranial aneurysms, dural arteriovenous malformations (AVM), stroke, intracranial atherosclerotic disease, dural arteriovenous fistulas (AVF)
13. Subject with an intracranial tumor
14. Subject with active or suspected acute or chronic uncontrolled infection
15. Subject had deep brain stimulation or a prior stereotactic ablation of the basal ganglia or thalamus
16. Patients with implanted objects in the skull or the brain
17. More than 30% of the skull area traversed by the sonication pathway is covered by scars, scalp disorders (e.g., eczema), or atrophy of the scalp
18. Subjects who have been administered botulinum toxins into the arm, neck, or face for 5 months prior to Baseline.
19. Subject has an overall Skull Density Ratio of less than 0.40 (±0.05) as calculated at screening
20. Subject is unable or willing to tolerate the required prolonged stationary supine position during Exablate procedure (approximately 2-3 hours)
21. Subject is currently participating in another clinical investigation with an active treatment arm
22. Subject is unable to communicate with the investigator and staff
23. Subject is considered to be a poor surgical or study candidate, which may include, but is not limited to the following: any medical, social, or psychological problem that could complicate the required procedures and evaluations of the study in the judgment of the investigator

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of Device and Procedure Related Adverse Events | 2 Years post treatment
  The cumulative sum of adverse events was followed through Year 2 of the study

SECONDARY OUTCOMES:
Tremor Motor Score - Clinical Rating Scale for Tremor (CRST) | Baseline,1 Month, 3 Months, 6 Months, 12 Months, 2 Years post treatment
  Sum of baseline and follow-up in upper extremity Tremor-Motor scores for the treated side is a sub-scale of Clinical Rating Scale for Tremor (CRST) Part A and Part B sum that was used to measure treated-side upper extremity tremor changes over time. Tremor-motor scores range from 0-32 points. Individual subject's scores at Baseline and Follow Up were calculated at baseline and follow-up visits averaged across subjects. Low scores are better (show improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Longsheng Pan Professor, MD, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No